CLINICAL TRIAL: NCT07267884
Title: Evaluation of the Effectiveness and Safety of Intra-Aortic Balloon Pump Insertion in Patients With Ventricular Septal Defect Following Myocardial Infarction During SCAI SHOCK Stage B: A Multicenter, Randomized, Open-Label, Parallel Controlled Study
Brief Title: IABP for MI-VSD Patients in SCAI SHOCK Stage B
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); The Second Hospital of Shandong University (Other); Jinan Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KYLL-202506-052-1
Record Dates: First submitted 2025-09-30; First posted 2025-12-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-09

CONDITIONS: Acute Myocardial Infarction (AMI); Ventricular Septal Defects (VSD)
Keywords: Intra-aortic balloon pump; acute myocardial infarction; ventricular septal defect; cardiogenic shock
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Open-Label, Parallel Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-CS-IABP group (Experimental): Immediate placement (within 8 hours) of an IABP followed by medication upon admission
  Interventions: Device: Insertion of IABP in SCAI SHOCK stage B
- Control group (No Intervention): Routine medication treatment upon admission. According to the current guidelines, patients will receive IABP insertion to maintain circulation when they progress to SCAI SHOCK stages C-E.

INTERVENTIONS:
Device: Insertion of IABP in SCAI SHOCK stage B — For patients in Early-CS-IABP group, IABP will be inserted within 8 hours after admission, along with medical treatment to maintain circulatory stability. Once the Department of Cardiovascular Surgery determines that a patient has surgical indications, he will be transferred to the surgery department for surgical septal repair.
  Arms: Early-CS-IABP group

SUMMARY:
Ventricular septal defect (MI-VSD) is a serious mechanical complication of acute myocardial infarction, with an extremely high mortality. Intra-aortic balloon pump (IABP) is still the most easily available mechanical assistive device for clinical management, and it has become a bridge to surgical repair.

IABP-SHOCK II trial is currently the largest randomized controlled trial (RCT) related to the use of IABP among patients with acute myocardial infarction (AMI) complicated by cardiogenic shock (CS), the trial found that IABP had a negative impact on 30-day, 1-year, and 6-year all-cause mortality. However, the trial included patients with typical cardiogenic shock (shock stages C-E, SCAI definition criteria), most of whom had severely inadequate microcirculatory perfusion, limiting the effectiveness of IABP treatment.

There is still no clinical study on the usage of IABP in MI-VSD patients with early-stage CS. The main objective of this study is to assess the correlation between the utilization of IABP and 30-day mortality rates among MI-VSD patients with early-stage CS. The investigators will also follow up on the long-term prognosis of these patients. The investigators will enroll multicenter patients with MI-VSD who are at the onset of cardiogenic shock (SCAI SHOCK stage B) to explore the impact of IABP support on the prognosis of these patients.

This prospective, multicenter, randomized, open-label, parallel-group controlled study will involve 100 participants who are diagnosed with MI-VSD complicated by SCAI SHOCK stage B in about 5 centers. After reviewing the inclusion criteria, participants will be randomized to two groups (Early-CS-IABP group and Control group) in a ratio of 1:1. The primary outcome is all-cause mortality within 30 days after MI-VSD. The investigators will also observe 6-month and 1-year all-cause mortality after MI-VSD.

The investigators speculated that IABP could significantly improve the clinical outcomes of patients with MI-VSD if it could be used in the early stage of cardiogenic shock.

DETAILED DESCRIPTION:
1. Background Ventricular septal rupture (MI-VSD) is a severe mechanical complication of acute myocardial infarction with an extremely high mortality rate. Previous studies have shown that MI-VSD occurs in 1% to 3% of patients with ST-segment elevation myocardial infarction (STEMI), and in patients with acute myocardial infarction complicated by cardiogenic shock (AMICS), the incidence of MI-VSD increases to 3.9% . The early and long-term prognosis for MI-VSD remains poor. A study found that the 30-day, 1-year, and 5-year mortality rates for patients with MI-VSD were 62%, 72%, and 95%, respectively, with the 30-day mortality rate for patients treated medically being 100%.

   Traditional shock stage criteria cannot accurately identify the pre-shock stage, thus failing to implement timely intervention measures to prevent hemodynamic deterioration. In 2022, the Society for Cardiovascular Angiography and Interventions (SCAI) proposed a shock stage classification system that divides shock into stage A to E, defined as at risk, beginning, classic, deteriorating, and extremis, providing a risk stratification for mortality in CS patients. According to this staging system, patients begin to exhibit significant hemodynamic disturbances and inadequate microcirculatory perfusion at SCAI SHOCK stage C, which is the typical cardiogenic shock stage.

   IABP-SHOCK II trial is currently the largest randomized controlled trial (RCT) related to the use of IABP among patients with AMICS. The trial found that IABP had a negative impact on all-cause mortality within 30 days, 1 year, and 6 years for AMICS patients. Therefore, the 2025 ACC/AHA/ACEP/NAEMSP/SCAI guidelines for the treatment of acute coronary syndrome (ACS) recommend against routine use of IABP as a standard supportive therapy in patients with AMICS. However, the trial included patients with typical cardiogenic shock (SCAI SHOCK stages C-E), most of whom had severely inadequate microcirculatory perfusion, limiting the effectiveness of IABP treatment. Patients with MI-VSD experienced rapid hemodynamic changes, and untreated ventricular septal perforation areas might further expand.

   Despite the current guideline downgrading the recommendation for routine use of IABP in patients with AMICS, it remains the most prevalent method utilized in clinical practice. According to the investigators' retrospective study based on MI-VSD patients who were admitted to Qilu Hospital of Shandong University from 2013 to 2024, the use of IABP could remarkably reduce the 30-day mortality and improve long-term prognosis in patients with early-stage cardiogenic shock (SCAI SHOCK stages A/B) at baseline, but did not improve outcomes in those with typical cardiogenic shock (SCAI SHOCK stages C-E).

   Significant differences between clinical practice and guidelines suggest that a specific population of MI-VSD patients may respond well to IABP support. This study aims to enroll multicenter patients with MI-VSD who are at the onset of cardiogenic shock (SCAI SHOCK stage B) to explore the impact of IABP support on the prognosis of these patients. This study include patients in shock stage B because they are at the beginning of AMICS and also a critical period for treatment.
2. Speculated conclusion The investigators speculated that IABP could significantly improve the clinical outcomes of patients with MI-VSD if it could be used in the early stage of cardiogenic shock.
3. Study Design 3.1 Design Prospective, multicenter, randomized, open-label, parallel-group controlled trial 3.2 Study Participant Grouping The grouping will be conducted using a central randomized complete random design. After reviewing the inclusion criteria, participants will be randomized to two groups in a ratio of 1:1. (1) Early-CS-IABP group: Immediate placement (within 8 hours) of an IABP followed by medication upon admission; (2) Control group: Routine medication treatment upon admission. According to the current guidelines, patients will receive IABP insertion to maintain circulation when they progress to SCAI SHOCK stages C-E. For patients with SCAI SHOCK stages C-E who have had IABP inserted, crossover to the early IABP group is not allowed, as they do not receive early intervention in stage B 3.3 Sample Size Based on the data from previous studies, assuming a 30-day all-cause mortality rate of 50% in the control group and an Early-CS-IABP group can reduce the mortality rate to 20%, with α=0.05 (two-sided) and β=0.1 (90% power), we calculate that at least 47 patients are needed in each group, totaling 94 patients. Considering 5% possible attrition and data loss, we aim to recruit a total of 100 participants.

3.4 Sample collection Whole blood specimen 10mL 4 Statistical Methods Statistical analysis will be conducted using SPSS and R. The population will be randomly divided into the IABP group and the control group. Baseline data and clinical outcomes of the study population will be compared for differences. Continuous variables will be analyzed for differences using T-tests, ANOVA, and nonparametric tests. Categorical variables will be analyzed using the chi-square test for statistical analysis. Kaplan-Meier survival curves will be used to estimate the 30-day cumulative mortality rates in the IABP group and the control group, and the Log-rank test will be used to compare the differences between the two groups. Subgroup analyses will be conducted to compare the association between early IABP implantation and 30-day all-cause mortality in different subgroups, and to analyze interactions. Secondary endpoints and safety endpoints will be evaluated using Fisher's exact test or the chi-square test for binary endpoint assessment, or the Mann-Whitney U test for quantitative endpoint assessment. The investigators will conduct Cox regression analysis to evaluate the impact of IABP implantation on 6-month and 1-year mortality. A p-value less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* Diagnosed with AMI based on electrocardiogram, cardiac troponin markers, etc.;
* Diagnosis of MI-VSD by echocardiography;
* Patients in stage B according to the SCAI SHOCK staging definition, meeting the following conditions: (1) Good mental status, (2) Warm limbs without cold and clammy feeling, (3) Killip class 2, with the beginning of wet rales at the lung bases, (4) Arterial blood gas lactate ≤ 2 mmol/L, (5) Normal renal function or mild renal impairment (creatinine increase less than 1.5 times baseline or eGFR decrease ≤ 50%), (6) No use of vasoactive drugs;
* Obtain informed consent.

Exclusion Criteria:

* Age > 75 years;
* Typical cardiogenic shock at admission (SCAI SHOCK stages C-E), any of the following: (1) altered mental status, (2) cold and clammy skin, (3) Killip class 3 or 4, (4) arterial blood gas lactate > 2 mmol/L, (5) severe liver and kidney function impairment, (6) use of vasoactive drugs to maintain blood pressure; or in shock risk period (stage A);
* Congenital heart disease with ventricular septal defect;
* Complications such as free wall rupture, papillary muscle dysfunction, etc.;
* Cardiopulmonary resuscitation > 30 minutes;
* Shock caused by other reasons (such as sepsis or hypovolemia);
* Patients with other serious accompanying diseases with an expected life span of less than 12 months;
* Aortic valve insufficiency more than grade II, aortic dissection or aneurysm cannot be ruled out;
* Difficulty in implanting IABP due to severe peripheral vascular disease;
* Pregnancy and lactation;
* Refusal to sign the informed consent form, or disagreement with IABP implantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality within 30 days after MI-VSD | From enrollment to the 30th day of MI-VSD

SECONDARY OUTCOMES:
Arterial blood gas lactate | The first 4 days after enrollment
Serum creatinine | The first 4 days after enrollment
C-reactive protein levels | The first 4 days after enrollment
Number of participants who progress to SCAI SHOCK stages C-E | 30 days after MI-VSD
  Participants meeting the following criteria will be considered to progress to SCAI SHOCK stages C-E: (1) altered mental status, (2) cold and clammy skin, (3) Killip class 3 or 4, (4) arterial blood gas lactate > 2 mmol/L, (5) severe liver and kidney function impairment, (6) use of vasoactive drugs to maintain blood pressure. In the case report form, participants with shock progression were recorded as "1" while those without progression were recorded as "0".
6-month all-cause mortality after MI-VSD | From enrollment to 6 months after MI-VSD
1-year all-cause mortality after MI-VSD | From enrollment to 1 year after MI-VSD

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Yang, Principal Investigator — Qilu Hospital of Shandong University, Department of Cardiology
Locations (1):
- Department of Cardiology, Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Demographic statistics Vital signs Current medical history Past medical history and accompanying diseases Examinations and laboratory tests results IABP usage information Other treatments Medication use Follow-up information
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 4 months and ending 2 years after the publication of results
Access Criteria: Access to the de-identified IPD will be granted to qualified researchers who provide a sound and methodologically valid research proposal.

REFERENCES:
- [Result] Leng L, Liu X, Song C, Ran X, Lin Z, Zhai C, Qin X, Cao G, Zhang C, Yang J. Intra-aortic balloon pump implantation in early-stage cardiogenic shock reduces 30-day mortality in patients with ventricular septal defect following myocardial infarction. Int J Cardiol. 2026 Jan 1;442:133895. doi: 10.1016/j.ijcard.2025.133895. Epub 2025 Sep 10. PMID 40939873
- [Result] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Result] Rao SV, O'Donoghue ML, Ruel M, Rab T, Tamis-Holland JE, Alexander JH, Baber U, Baker H, Cohen MG, Cruz-Ruiz M, Davis LL, de Lemos JA, DeWald TA, Elgendy IY, Feldman DN, Goyal A, Isiadinso I, Menon V, Morrow DA, Mukherjee D, Platz E, Promes SB, Sandner S, Sandoval Y, Schunder R, Shah B, Stopyra JP, Talbot AW, Taub PR, Williams MS. 2025 ACC/AHA/ACEP/NAEMSP/SCAI Guideline for the Management of Patients With Acute Coronary Syndromes: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2025 Apr;151(13):e771-e862. doi: 10.1161/CIR.0000000000001309. Epub 2025 Feb 27. PMID 40014670
- [Result] Thiele H, Zeymer U, Neumann FJ, Ferenc M, Olbrich HG, Hausleiter J, Richardt G, Hennersdorf M, Empen K, Fuernau G, Desch S, Eitel I, Hambrecht R, Fuhrmann J, Bohm M, Ebelt H, Schneider S, Schuler G, Werdan K; IABP-SHOCK II Trial Investigators. Intraaortic balloon support for myocardial infarction with cardiogenic shock. N Engl J Med. 2012 Oct 4;367(14):1287-96. doi: 10.1056/NEJMoa1208410. Epub 2012 Aug 26. PMID 22920912
- [Result] Naidu SS, Baran DA, Jentzer JC, Hollenberg SM, van Diepen S, Basir MB, Grines CL, Diercks DB, Hall S, Kapur NK, Kent W, Rao SV, Samsky MD, Thiele H, Truesdell AG, Henry TD. SCAI SHOCK Stage Classification Expert Consensus Update: A Review and Incorporation of Validation Studies: This statement was endorsed by the American College of Cardiology (ACC), American College of Emergency Physicians (ACEP), American Heart Association (AHA), European Society of Cardiology (ESC) Association for Acute Cardiovascular Care (ACVC), International Society for Heart and Lung Transplantation (ISHLT), Society of Critical Care Medicine (SCCM), and Society of Thoracic Surgeons (STS) in December 2021. J Am Coll Cardiol. 2022 Mar 8;79(9):933-946. doi: 10.1016/j.jacc.2022.01.018. Epub 2022 Jan 31. No abstract available. PMID 35115207
- [Result] Poulsen SH, Praestholm M, Munk K, Wierup P, Egeblad H, Nielsen-Kudsk JE. Ventricular septal rupture complicating acute myocardial infarction: clinical characteristics and contemporary outcome. Ann Thorac Surg. 2008 May;85(5):1591-6. doi: 10.1016/j.athoracsur.2008.01.010. PMID 18442545
- [Result] Khan MY, Waqar T, Qaisrani PG, Khan AZ, Khan MS, Zaman H, Jalal A. Surgical Repair of post-infarction ventricular septal rupture: Determinants of operative mortality and survival outcome analysis. Pak J Med Sci. 2018 Jan-Feb;34(1):20-26. doi: 10.12669/pjms.341.13906. PMID 29643872
- [Result] Figueras J, Alcalde O, Barrabes JA, Serra V, Alguersuari J, Cortadellas J, Lidon RM. Changes in hospital mortality rates in 425 patients with acute ST-elevation myocardial infarction and cardiac rupture over a 30-year period. Circulation. 2008 Dec 16;118(25):2783-9. doi: 10.1161/CIRCULATIONAHA.108.776690. Epub 2008 Dec 8. PMID 19064683
- [Result] Matteucci M, Ronco D, Corazzari C, Fina D, Jiritano F, Meani P, Kowalewski M, Beghi C, Lorusso R. Surgical Repair of Postinfarction Ventricular Septal Rupture: Systematic Review and Meta-Analysis. Ann Thorac Surg. 2021 Jul;112(1):326-337. doi: 10.1016/j.athoracsur.2020.08.050. Epub 2020 Nov 4. PMID 33157063